CLINICAL TRIAL: NCT06699901
Title: Antibiotic Concentrations After MassivE Transfusion (ACME) Study
Brief Title: Antibiotic Concentrations After MassivE Transfusion Study
Acronym: ACME
Status: Recruiting | Type: Observational
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); The Metis Foundation (Other); University of Colorado Health (Other)
Responsible Party: Principal Investigator, Steven Schauer, PRINCIPAL INVESTIGATOR, Brooke Army Medical Center
Other Study IDs: 23-2559; HT9425-23-1-1074 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2024-10-31; First posted 2024-11-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Adverse Effects in the Therapeutic Use of Other and Unspecified Agents Affecting Blood Constituents
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples are retained, with no potential for DNA extraction from any retained samples. This study requires 1mL of whole blood to be collected in standard clinical sample tubes with anticoagulants and stored on ice or in a refrigerator (4°C) temporarily (total research sample volume from all timepoints = 6mL). As soon as feasible, the samples will be centrifuged for 10 minutes at 3000G, and the plasma will be removed and frozen at -80°C by a study team member. No other samples will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Patients who ideally receive no blood but may be included if they receive up to 2 units of transfused blood.
  Interventions: Other: Control Group
- Massive Transfusion Group: Patients who receive at least 3 units of blood.
  Interventions: Other: Massive Transfusion Group

INTERVENTIONS:
Other: Massive Transfusion Group — This group includes trauma patients who receive a massive transfusion, defined as the transfusion of at least 3 units of blood. Blood samples are collected at six specific timepoints following the administration of antibiotics to analyze plasma antibiotic concentrations. Existing clinical draws will be used whenever possible to minimize additional venipunctures, with a maximum of two dedicated research-only draws allowed if necessary. Data analysis will assess the impact of large blood transfusions on antibiotic pharmacokinetics over time, adjusting for factors such as kidney function.
  Groups: Massive Transfusion Group
Other: Control Group — This group consists of trauma patients who receive minimal or no blood transfusions (up to 2 units of blood). Blood samples are also collected at six designated timepoints after antibiotic administration to measure plasma antibiotic concentrations. As with the massive transfusion group, clinical draws will be coordinated whenever possible to obtain research samples, with a maximum of two dedicated research-only draws if needed. Data analysis will compare antibiotic concentration trends in this group with those in the massive transfusion group to understand the effects of blood transfusion volume on antibiotic pharmacokinetics.
  Groups: Control Group

SUMMARY:
Combat and civilian trauma frequently result in open wounds that are at risk for infection. Data from the Department of Defense Trauma Registry demonstrate that 74% of combat trauma casualties have an open wound. The Committee on Tactical Combat Casualty Care, the Prolonged Field Care Working Group, and the Joint Trauma System clinical practice guidelines recommend antibiotic prophylaxis for open wounds after trauma. The civilian setting has similar risks of open wound infection after trauma. In parallel, current practice guidelines recommend the aggressive use of balanced blood products during resuscitation. It remains unclear how the replacement of blood after hemorrhage through transfusion may affect antibiotic concentrations. Data is necessary to better understand this relationship to enhance wound prophylaxis antibiotic dosing, particularly in severely wounded casualties who receive blood products during massive transfusions. It remains unclear how these resuscitation methods may alter pharmacokinetics. The investigators hypothesize that drug concentrations decrease in direct relation to the amount of blood transfused during low-volume, massive, and supermassive transfusion after trauma compared to patients who receive no blood products. The investigators seek to understand the relationship between drug concentrations and blood product administration using a non-compartmentalized model in the setting of hemorrhage. Specifically, they will (1) obtain drug concentrations at regular intervals during the first 12-18 hours after administration of antibiotics, (2) determine how much blood products and fluids are transfused during the 12 hours prior to antibiotic and 24 hours post-administration, and (3) perform data modeling to understand the relationship between blood transfusions and drug concentrations to inform data-driven dosing models. Liquid chromatography methods will be developed to measure drug concentrations. The investigators will conduct a prospective, multicenter study at two large trauma centers - Brooke Army Medical Center and the University of Colorado Hospital. They will seek to enroll any participant who is hospitalized or anticipated hospital admission for acute trauma and receives an antibiotic on the study list during their index hospitalization. They will then model the drug levels against the amount of blood and fluid infused to create an understanding of the pharmacokinetics of antibiotic wound prophylaxis.

DETAILED DESCRIPTION:
This observational study evaluates the impact of blood transfusion volume on antibiotic plasma concentration in trauma patients. Participants who meet trauma criteria in the ED and receive specified antibiotics during their hospitalization are identified through trauma alerts, clinical engagement, and pharmacist involvement. A convenience sample will be enrolled, aiming for a 1:2 ratio of transfused patients to controls. Blood samples (1mL per timepoint) will be taken at six intervals post-antibiotic infusion, often aligning with clinical draws to minimize additional venipunctures. Samples will be processed, stored, and shipped to the USAISR lab for analysis, with data entered into REDCap for de-identified storage and future analysis. Statistical methods include descriptive and inferential statistics, regression modeling, ANOVA, and regression analysis to assess concentration differences by transfusion status and volume. Data is secured under HIPAA regulations, and minimal additional risk qualifies the study for a waiver of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Receives ampicillin/sulbactam, cefazolin, cefepime, ceftriaxone, clindamycin, ertapenem, levofloxacin, metronidazole or pipercillin/tazobactam at any dose
* Hospitalized or anticipated hospital admission

Exclusion Criteria:

* Received the same antibiotic within the past 5 half-lives of the drug (e.g. received the same antibiotic during a recent interval)
* <18 years of age
* Known pregnancy
* Known Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients brought to study sites who receive an antibiotic during their index hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Amount of drug concentrations within first 18 hours. | From initial enrollment until 30 days after.
  Obtain drug concentrations at regular intervals during the first 18 hours after antibiotic administration.

SECONDARY OUTCOMES:
Total volume of blood products within 24 hours. | From initial enrollment until 30 days after.
  Determine the total volume of blood products and fluids transfused during the first 24 hours after antibiotic administration.
Correlation Between Blood Transfusion Volume and Drug Concentration Levels | Through study completion, an average of 3 years.
  Assess the correlation between the volume of blood transfusions administered and resulting drug concentration levels. Blood transfusion volume will be recorded in milliliters (mL), and drug concentration levels will be measured in nanograms per milliliter (ng/mL) using Liquid Chromatography/Tandem Mass Spectrometry Methods (LC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Rizzo, MD, Principal Investigator — Brooke Army Medical Center
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Brooke Army Medical Center, Fort Sam Houston, Texas

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not authorized without a written agreement with the Defense Health Agency.

REFERENCES:
- [Background] Burbank KM, Schauer SG, De Lorenzo RA, Wenke JC. Early application of topical antibiotic powder in open-fracture wounds: A strategy to prevent biofilm formation and infections. OTA Int. 2020 Oct 12;3(4):e091. doi: 10.1097/OI9.0000000000000091. eCollection 2020 Dec. PMID 33937714
- [Background] Schauer SG, Naylor JF, Ahmed YM, Maddry JK, April MD. Prehospital Combat Wound Medication Pack Administration in Iraq and Afghanistan: A Department of Defense Trauma Registry Analysis. J Spec Oper Med. 2020 Fall;20(3):76-80. doi: 10.55460/X4E8-NNXE. PMID 32969008
- [Background] Eastridge BJ, Hardin M, Cantrell J, Oetjen-Gerdes L, Zubko T, Mallak C, Wade CE, Simmons J, Mace J, Mabry R, Bolenbaucher R, Blackbourne LH. Died of wounds on the battlefield: causation and implications for improving combat casualty care. J Trauma. 2011 Jul;71(1 Suppl):S4-8. doi: 10.1097/TA.0b013e318221147b. PMID 21795876
- [Background] Schauer SG, Naylor JF, Fisher AD, April MD, Hill R, Mdaki K, Becker TE, Bebarta VS, Bynum J. An Analysis of 13 Years of Prehospital Combat Casualty Care: Implications for Maintaining a Ready Medical Force. Prehosp Emerg Care. 2022 May-Jun;26(3):370-379. doi: 10.1080/10903127.2021.1907491. Epub 2021 Apr 16. PMID 33760684
- [Background] Fisher AD, Lavender JS, April MD, Hill R, Bynum J, Schauer SG. A Descriptive Analysis of Supermassive Transfusion Recipients Among US and Coalition Forces During Combat Operations in Afghanistan and Iraq. Mil Med. 2023 May 16;188(5-6):e1022-e1027. doi: 10.1093/milmed/usab455. PMID 34741519
- [Background] Shackelford SA, Del Junco DJ, Powell-Dunford N, Mazuchowski EL, Howard JT, Kotwal RS, Gurney J, Butler FK Jr, Gross K, Stockinger ZT. Association of Prehospital Blood Product Transfusion During Medical Evacuation of Combat Casualties in Afghanistan With Acute and 30-Day Survival. JAMA. 2017 Oct 24;318(16):1581-1591. doi: 10.1001/jama.2017.15097. PMID 29067429
- [Background] Eastridge BJ, Mabry RL, Seguin P, Cantrell J, Tops T, Uribe P, Mallett O, Zubko T, Oetjen-Gerdes L, Rasmussen TE, Butler FK, Kotwal RS, Holcomb JB, Wade C, Champion H, Lawnick M, Moores L, Blackbourne LH. Death on the battlefield (2001-2011): implications for the future of combat casualty care. J Trauma Acute Care Surg. 2012 Dec;73(6 Suppl 5):S431-7. doi: 10.1097/TA.0b013e3182755dcc. PMID 23192066

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT06699901/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT06699901/ICF_001.pdf